CLINICAL TRIAL: NCT01623154
Title: A Prospective, Multi-Center, Open-Label Study to Compare the POCone® With the UBiT®-IR300 in Measurement of 13CO2/12CO2 Ratio in Breath Samples Collected From Pediatric Subjects Ages 3 to 17 Years With Upper Gastrointestinal Signs and Symptoms
Brief Title: POCone-UBiT-IR300 Pediatric Comparison Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UBT-1l-202
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
Keywords: Helicobacter pylori

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BreathTek UBT (Other): Comparison of Urea hydrolysis rate (UHR) values derived from Delta over Baseline (DOB)values obtained from the POCone and UBiT-IR300
  Interventions: Other: Pranactin citric solution

INTERVENTIONS:
Other: Pranactin citric solution — All patients were required to drink the pranactic citric solution to diagnose H.pylori.

SUMMARY:
The purpose of this study is to compare between the POCone® to the UBiT®-IR300 in measuring 13CO2/12CO2 ratio in breath samples when used together with the BreathTek® UBT (urea breath test) Kit and the pUHR-CA web-based software program in identifying H. pylori infection in pediatric subjects.

DETAILED DESCRIPTION:
The same patients will be tested on both the POCone® and UBiT®-IR300. If the patients test positive for H. pylori, they will be given eradication medication and brought back in for a re-test.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ages 3 to 1711/12 years.
2. Subject with upper gastrointestinal signs and symptoms (e.g., abdominal pain/discomfort, bloating, nausea, or vomiting, etc.)
3. Subject and/or parent/legal guardian is capable of giving assent or consent.
4. Subject is able to complete the urea breath test by investigator's assessment.

Exclusion Criteria:

1. Subject is hypersensitive to mannitol, citric acid and/or aspartame.
2. Previous diagnosis of phenylketonuria (PKU.
3. Subject with difficulty swallowing or who may be at high risk for aspiration due to medical or physical conditions.
4. Subjects with ongoing respiratory conditions or on bronchodilators that may compromise the collection of breath samples.
5. Subjects with severe chronic illness (e.g., Crohn's disease, leukemia, kidney diseases, etc.)
6. Administration of bismuth preparations (e.g., Pepto-Bismol®) at anytime within 14 days prior to the testing.
7. Administration of antibiotics (e.g., amoxicillin, tetracycline, metronidazole, clarithromycin, azithromycin, etc.) therapy at anytime within 14 days prior to the testing.
8. Administration of proton pump inhibitors (PPI; e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, pantoprazole, etc.) at anytime within 14 days prior to the testing.
9. Administration of Histamine H2 receptor antagonist (H2RA; e.g., ranitidine, cimetidine, famotidine, nizatidine, etc.) at anytime within 24 hours prior to the testing.
10. Treatment for eradication of H pylori within 28 days before testing or retesting.
11. Participation in a drug or device study within 30 days of testing

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami Pediatric Gastroenterology, Miami, Florida
  - University of Texas School of Public Health, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Urea Hydrolysis Rate (UHR): Urea hydrolysis rate (UHR) values derived from Delta over Baseline (DOB)values obtained from the POCone and UBiT -IR300
  Same patients will be tested on both the POCone and UBiT-IR300
Period: Overall Study
Arm/Group | Urea Hydrolysis Rate (UHR)
Started | 99
Available for Analysis | 95
Completed | 95
Not Completed | 4
Not completed — Did not drink Pranactin Citric | 4

BASELINE CHARACTERISTICS:
Population: 95 evaluable subjects for initial diagnosis- each patient received the BreathTek UBT test. Collected breath samples were analyzed on both the UBiT-IR300 and the POC-one.
Groups:
- BreathTek UBT: Comparison of urea hydrolysis rate (UHR) values derived from Delta over Baseline (DOB)values obtained from the POCone and UBiT-IR300. UBiT-IR300 is the FDA approved device.
Arm/Group | BreathTek UBT
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants] — Must drink the entire content of test solution and receive initial BreathTek UBT of both the UBiT-IR300 and the POC One
  Participants
    <=18 years | 95
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.5 [3.4 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 41
Region of Enrollment [Number; unit: Number of Participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between POCone and UBiT-IR300.
Description: The study end-points are UHR values derived from DOB (delta over baseline) values obtained from the POCone and UBiT-IR300 (UHRP and UHRU, respectively) at Baseline and Post-Dose. Same patients will be tested on both the POCone and UBiT-IR300.
  Subjects fasted for at least 1 hr prior test. Each patient provided breath samples in 3 blue (Baseline) breath bags-labeled "A" "B" "C". Subjects were given Pranactin-Citric solution (4oz) to drink, waited 15 min and collected 3 pink (post-dose) bags which were paired with the baseline bags in no particular order. Each pair was tested on both machines. The first two available pairs of UHR values were used for data analysis. The 3rd pair was used only if one of the first two samples did not produce a valid test result.
  DOB values were generated by the two instruments for each Baseline and Post Dose pair. UHR values were claculated based on the DOB values and the subject's anthropometric variables (age, gender, ehight and body weight).
Time Frame: Baseline, Post Dose (15 min)
Population: Evaluable patients must drink all of the Pranactin-citric solution. Though all three sets of bags were analysed, the first two sets of valid values were used for analysis, regardless of the set designation (A, B or C). The values of individual sets (A, B or C) were not analyzed.
Measure: Number (95% Confidence Interval)
Groups:
- Urea Hydrolysis Rate (UHR) Values: Urea hydrolysis rate (UHR) values derived from Delta over Baseline (DOB)values obtained from the POCone compared to the the approved device, UBiT-IR300. Three regression analyses completed (Deming, Passing-Bablok and Regular regression).
Arm/Group | Urea Hydrolysis Rate (UHR) Values
Number analyzed (Participants) | 95
Value
  Deming Regression Analysis | 0.990 [0.987 to 0.993]
  Passing-Bablok Regression Analysis | 0.995 [0.990 to 1.00]
  Regular Regression Analysis | 0.990 [0.987 to 0.993]
Statistical Analysis 1: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — While 40 subjects is the min req by the NCCLS guideline on method comparison (EP9-A2), we proposed to enroll a min of 60 evaluable pediatric subjects (max of 80) with at least 20 of them having a UHR value of ≥ 10.0µg/min. The expected # of positive cases is 20-30% of the subjects enrolled, we anticipated that 80 eval subj would give approximately 20 subj with a pos UHR value. The anticipated % pos/neg agreement between the 2 instruments is 95% bases on data from the adult population; Deming Regression — 95% confidence interval is used instead of p-value; Analyses to determine the comparability between UHR & DOB values from the 2 instruments included Deming, Passing-Bablok and regular regressions; Slope = 0.99, 95% CI 2-sided [0.987 to 0.993] — 95% confidence interval is used instead of p-value
Statistical Analysis 2: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Deming Regression; [statistical method as in outcome 1, analysis 1]; Intercept = -.04, 95% CI 2-sided [-0.25 to 0.17] — 95% confidence interval is used instead of p-value
Statistical Analysis 3: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = 0.990, 95% CI 2-sided [0.987 to 0.993] — 95% confidence interval is used instead of p-value
Statistical Analysis 4: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Linear; [statistical method as in outcome 1, analysis 1]; Intercept = -0.03, 95% CI 2-sided [-0.24 to 0.18] — 95% confidence interval is used instead of p-value
Statistical Analysis 5: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Passing-Bablock; [statistical method as in outcome 1, analysis 1]; Slope = 0.995, 95% CI 2-sided [0.990 to 1.000] — 95% confidence interval is used instead of p-value
Statistical Analysis 6: Comparison: Urea Hydrolysis Rate (UHR) Values; While 40 subjects is the min req by the NCCLS guideline on method comparison (EP9-A2), we proposed to enroll a min of 60 evaluable pediatric subjects (max of 80) with at least 20 of them having a UHR value of ≥ 10.0µg/min. The expected # of positive cases is 20-30% of the subjects enrolled, we anticipated that 80 eval subj would give approximately 20 subj with a pos UHR value. The anticipated % pos/neg agreement between the 2 instruments is 95% bases on data from the adult population; Test type: Non-Inferiority or Equivalence — Analyses to determine the comparability between UHR & DOB values from the 2 instruments included Deming, Passing-Bablok and regular regressions; Passing-Bablok; [statistical method as in outcome 1, analysis 1]; Intercept = -0.04, 95% CI 2-sided [-0.30 to 0.01] — 95% confidence interval is used instead of p-value
Statistical Analysis 7: Comparison: Urea Hydrolysis Rate (UHR) Values; Comparison of UHR Values obtained by UBit-IR300 and POCone were used to identify participants' H.pylori infection status. Participants with UHR value ≥ 10.0μg/min were considered positive for H.Pylori; Test type: Non-Inferiority or Equivalence — Described previously; Relative Sensitivity, % = 100, 95% CI 2-sided [85.8 to 100] — 95% confidence interval is used instead of p-value
Statistical Analysis 8: Comparison: Urea Hydrolysis Rate (UHR) Values; Test type: Non-Inferiority or Equivalence — Provided previously; Relative Specificity, % = 100, 95% CI 2-sided [94.9 to 100] — 95% confidence interval is used instead of p-value

2. Other Pre Specified Outcome: Number of Participants Tested Positive/Negative for H. Pylori
Description: Qualified subjects from clinical sites underwent a standard urea breath test using the BreathTek UBT Kit. Breath samples were analyzed using both the POCone and the UBiT-IR300. DOB values from these two infrared spectrophotometers were converted to respective UHR values using pUHR-CA. The paired UHR values from each subject were evaluated for agreement.
  UHR values of >10 µg/min were considered positive for H. pylori and UHR values of <10 µg/min were considered negative for H. pylori.
Time Frame: Single Study Visit (1 hour of testing)
Population: 95 evaluable subjects for initial diagnosis - each patient received the BreathTek UBT test. Collected breath samples were analyzed on both the UBiT-IR300 and the POC-one.
Measure: Number; unit: Participants
Groups:
- UBiT-IR300: This is the FDA approved device.
- POCone: This is the device being tested and compared to the FDA approved device.
Arm/Group | UBiT-IR300 | POCone
Number analyzed (Participants) | 95 | 95
Participants
  Positive for H.pylori | 24 | 24
  Negative for H. pylori | 71 | 71

ADVERSE EVENTS:
Description: At each visit, each subject received 1 administration of Pranactin Citric (4 oz of solution in water). This was the only component with patient contact. Hence, there is only one arm for adverse events evaluation.
Groups:
- Pranactin Citric Solution: At each visit, each subject provided baseline breath samples by exhaling into the mouthpiece of the 3 Baseline bags (Blue bags, labeled A,B, C according to collection order), received one 4 oz administration of Pranctin Citric solution (mixed in water, drink using a straw), waited 15 minutes and provided the Post-Dose breath samples (Pink bags, labeled A, B, C). The Blue and Pink bags were paired and tested in no particular order on each instrument. The subjects who tested positive for H.pylori underwent a second set of tests 28 days after completion of eradication therapy.
Arm/Group | Pranactin Citric Solution
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 4/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pranactin Citric Solution (N=99)
Headache (Nervous system disorders) | 2 (2) — Headache
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — cough
Dry Mouth (Gastrointestinal disorders) | 1 (1) — Dry Mouth
Acute Upper Respiratory Infection (Infections and infestations) | 1 (1) — Acute Upper Respiratory Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Central/Principal Investigator may publish the results of the study. However, at least 60 days prior to submitting to a publisher or a public presentation, a copy of the manuscript will be provided to the Sponsor for review. PI understands and agrees that as such, participation in the study involves a commitment to publish the data from the study in a cooperative publication prior to publication or oral presentation of efficacy/safety results on an individual basis.